CLINICAL TRIAL: NCT04521179
Title: A Phase II, Open-Label, Multi-Center Study to Evaluate Efficacy, Safety and Tolerability of KN026 in Combination With KN046 in Patients With Locally Advanced Unresectable or Metastatic HER2-positive Solid Tumors
Brief Title: Study of KN026 Combined With KN046 in Patients With Locally Advanced HER2-positive Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Collaborators: Peking University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KN026-203
Record Dates: First submitted 2020-08-18; First posted 2020-08-20 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-05

CONDITIONS: HER2-positive Solid Tumors
Keywords: KN026 and KN046; HER2-Positive Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KN026 combined with KN046 (Experimental): KN026 combination therapy
  Interventions: Drug: KN026 combination

INTERVENTIONS:
Drug: KN026 combination — 30 mg/kg Q3W KN026+ 5 mg/kg Q3W KN046
  Other Names: IO therapy

SUMMARY:
This is an open-label, phase II，multi-center study to evaluate the efficacy, safety and tolerability of KN026 in combination with KN046 in subjects with HER2-positive solid tumors.

DETAILED DESCRIPTION:
KN026 is an anti-HER2 bispecific antibody that can simultaneously bind two non-overlapping epitopes of HER2, leading to a dual HER2 signal blockade.KN046 is a PD-L1 - CTLA-4 bispecific antibody. The study composes of two stages. The first stage plans to enroll HER2-positive solid tumors. All subjects will be treated with KN026 at 30 mg/kg Q3W in combination with KN046 at 5 mg/kg Q3W at the first stage.A SMC meeting will decide whether to proceed to the nest stage.

ELIGIBILITY:
Inclusion Criteria:

* The subject can understand the informed consent, voluntarily participate and sign the informed consent ;
* Subjects are older than or equal to 18 years old and younger than or equal to 75 years old on the day of signing the informed consent；
* Histologically or cytologically confirmed, metastatic or locally advanced unresectable HER2-positive solid tumors;
* Prior antitumor therapy needs to meet the following conditions:

Her2-positive GC/GEJ: has not received prior systemic treatment for metastatic or locally advanced unresectable GC/GEJ, or has received prior systemic treatment≥1 line of systemic treatment with disease progression, front-line systemic treatment includes at least platinum or fluorouracil based chemotherapy with or without trastuzumab; Subjects who relapsed within 6 months after the end of neoadjuvant/adjuvant chemotherapy were considered as line 1 treatment failure; Her2-positive BC: prior treatment with ≥1 line of HER2-targeted therapy for metastatic disease and disease progression; Subjects who relapsed within 12 months after the end of neoadjuvant/adjuvant chemotherapy were considered as line 1 treatment failure; Other HER2-positive solid tumors: previous ≥1 line of systemic therapy for metastatic or locally advanced unresectable tumors with disease progression, no clear standard therapy for prolongation of survival, or after subjects rejected 1 line of systemic therapy; Frontline systemic therapy for ovarian and cervical cancer includes at least platinum-based (cisplatin or carboplatin) chemotherapy; Frontline systemic therapy for ESCC and mCRC includes at least platinum combined with fluorouracil or tax-based chemotherapy; MCRC requires ≥2 lines of systemic therapy for metastatic or locally advanced unresectable tumors and disease progression; Subjects who relapsed within 6 months after completion of neoadjuvant/adjuvant platinum-containing chemotherapy Line 1 treatment failure;

* At least 1 measurable lesion at baseline according to RECIST1.1 criteria；
* ECOG score 0 or 1;
* Left ventricular ejection fraction (LVEF) ≥ 50% at baseline as determined by either ECHO (preferred) or MUGA;
* Liver function met the following criteria within 7 days prior to initial administration:

Total bilirubin ≤1.0x ULN (Gilbert's syndrome, or total bilirubin ≤1.5x ULN in liver metastases); Aminotransferase (ALT/AST) ≤1.5x ULN (liver metastatic subjects ≤3xULN); -Renal function within 7 days prior to initial administration: serum creatinine ≤1.5x ULN and serum creatinine clearance ≥60mL/min (according to Cockcroft-Gault Formula calculation);

-Bone marrow function met the following criteria within 7 days prior to initial administration: Hemoglobin ≥90 g/L; Neutrophil absolute count ≥1.5 x 109/L; Platelet count ≥100x 109/L; INR or PT≤1.5x ULN, and aPTT≤ 1.5x ULN;

* TSH normal range： If TSH is abnormal, total or free T3 and free T4 should be in the normal range
* Life expectancy >3 months;
* Fertile female subjects or fertile male subjects with a partner agreed to use hepa beginning 7 days prior to the first dose pregnancy continued until 24 weeks after drug withdrawal. Fertile female subjects must have a negative serum pregnancy test within 7 days prior to first dosing;
* The subjects are able and willing to follow the visits, treatment plans, laboratory tests, and other study-related procedures specified in the study protocol

Exclusion Criteria:

* Untreated active brain metastasis or leptomeningeal metastasis;
* Historyof Left ventricular ejection fraction (LVEF) decline to < 45% or absolute decrease for > 15% during the treatment course from prior HER2-targeted therapy;
* Previous cumulative doses of anthracycline exceeded doxorubicin or liposomal doxorubicin >320mg/m2 or equivalent doses of other anthracyclines;
* Has received other anti-tumor treatment or an investigational drug within 28 days or 5 half-lives prior(whichever is shorter, but at least 2 weeks) to the first trial treatment;
* Major surgery (transabdominal, transthoracic, etc.) within 28 days prior to initial administration; Diagnostic puncture or peripheral vascular is not included pathway replacement)
* Radical radiotherapy within 3 months prior to initial administration; Palliative radiotherapy is allowed 2 weeks before administration, and the dose of radiotherapy is in line with local palliative the diagnosis and treatment standard of sexual therapy and the coverage of radiotherapy is less than 30% of the bone marrow region;
* Prior treatment with immune checkpoint blockers or T cell costimulators;
* Systemic corticosteroid or immunosuppressant therapy is required for 7 consecutive days within 14 days of initial dosing
* Received live vaccines (including attenuated live vaccines) within 28 days of initial administration;
* Have interstitial lung disease or a history of non-infectious pneumonia requiring oral or intravenous glucocorticoid treatment;
* Have a past or current autoimmune disease;
* Other malignant tumors occurred within 5 years prior to initial administration;
* With uncontrolled comorbidities;
* Toxicity from previous antitumor therapy did not return to CTCAE grade ≤1 (NCI-CTCAEV 5.0) or baseline levels;
* Prior allo-HSCT or solid organ transplant;
* History of allergic reaction, hypersensitivity reaction and intolerance to antibody drugs; Prior allergic reaction to medication ;
* Pregnant or nursing females;
* Other medical conditions that at the discretion of investigator interfere with the requirements of the trial in terms of safety or efficacy evaluation, or treatment compliance;
* BMI less than 18.5kg/m2 or weight loss ≥10% within 2 months prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR ) | Throughout the duration of the study; up to 2 years
  Objective response rate as assessed by the investigator according to RECIST 1.1 criteria
Duration of response (DOR) | Throughout the duration of the study; up to 2 years
  Duration of response (DOR) as assessed by the investigator according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
Progression free survival (PFS) rates | 6 months and 12 months
  Progression free survival (PFS) rates
Clinical benefit rate (CBR) | CBR calculated as the proportion of subjects with best overall response of CR, PR, or SD ≥24 weeks
  Clinical benefit rate
Overall survival (OS) | 6 months and 12 months
  Overall survival (OS) rates

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, professor, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liao JY, Wang J, Li H, Liu Z, Tian Z, Lv X, Peng J, Song C, Liu J. Longitudinal tissue analysis reveals microenvironmental changes correlate with combined immunotherapy and targeted therapy response in metastatic breast cancer. J Immunother Cancer. 2025 Oct 5;13(10):e012629. doi: 10.1136/jitc-2025-012629. PMID 41052881